CLINICAL TRIAL: NCT05334771
Title: Early Detection of Endolymphatic Hydrops in Hypothyroid Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Ali Abdelazeem Mohamed, princible invistigator, Assiut University
Other Study IDs: Hypothyroidism
Record Dates: First submitted 2022-03-11; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Acoustic Impedance Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Dual band pure tune audiometer — Orbiter 922 Tympanometry
  Other Names: Impedance audiometry

SUMMARY:
Early detection of endolymphatic hydrops in hypothyroid patients Study outcome of medical treatment for hypothyroid patients

DETAILED DESCRIPTION:
Endolymphatic hydrops is acommon inner ear dysfunction. This term often used with meniere's disease and meniere's syndrome. However meniere's is idiopathic by definition where as it can occur secondary to various processes interfering with normal production or absorption of endolymph. Histopathologically, endolymphatic hydrops is seen initially in the cochlear duct and the saccule; with the progression of the disease, subsequent affection of the utricle and semicircular canals (SCC) occur . Vascular alterations, genetic predisposition, hormonal disorders and nutritional and psychological factors might contribute to the genesis of hydrops . Serum antibodies against internal ear antigens and circulating immunocomplexes as well as apositive response to steroid treatment have been reported. Furthermore, MD patients present some features of immune diseases, such as hereditary predisposition, apositive family history for the disease and hypothetic association with certain human leucocyte antigen loci (Cw7, A1, B8) .

The thyroid gland has crucial functions to regulate the endocrine systems through the hypothalamic-pituitarythyroid axis and affect organ-specific such as as Addison's disease and type 1 diabetes mellitus or non-organ-specific such as rheumatoid arthritis and systemic lupus erythematosus .

Ménière's disease is clinically diagnosed by recurrent vertigo attacks combined with cochlear symptoms of primarily low- or mid-frequency sensorineural hearing loss, tinnitus, or ear fullness . The incidence of Ménière's disease varies according to the ethnic population, which is estimated to be about 13-200 person-years . The peak age of onset of Ménière's disease has been reported to be about 40-60 years . The sudden surge of endolymphatic flow, which shifts from the pars inferior (cochlea) to the pars superior (utricle and semicircular canals), stimulates the vestibular hair cells in the cristae of the semicircular canals and may induce vertigo attack in patients with Ménière's disease. However, the pathophysiologic causes for the increase of endolymphatic flow are not understood and are thought to be multifactorial, including abnormal immune response and metabolic endocrine dysfunctions, such as hypothyroidism. Previous studies have suggested the association of hypothyroidism with Ménière's disease . Many studies reported high incidence of thyroid dysfunction in Ménière's disease.

The possible association between (autoimmune) thyroid disease and MD has been postulated for more than 30 years, but it is still controversial. Pulec and House first reported that 3% of patients with MD had a positive history for hyperthyroidism, and Powers et al. found a much higher prevalence of association between MD and hypothyroidism. However, at the beginning of the 1980s, arelationship between altered thyroid function and MD was actually excluded by Kinney and by Meyerhoff et al. , while Evans et al. showed subsequently that 17% of sera from MD patients contained positive anti-thyroidmicrosome antibody titres.

The assessment of patients with Ménière's disease can be challenging. VEMP findings in Meniere's patients varies based on the acuteness and stage of the disease. ~50% of patients with Meniere's disease have asymmetric CVEMP responses, indicating differences in the saccular function (returns to normal in ~50%). Recent reports show different frequency tuning in CVEMP thresholds for 250 Hz - 1 kHz stimuli in patients with endolymphatic hydrops. Some patients show the same pattern in the unaffected ear, perhaps indicating delayed endolymphatic hydrops. 40% of Meniere's patients show improvement in cVEMP amplitude following the administration of furosemide (Seo et al, 2003).

VEMP is aneurophysiological assisment technique to evaluate the patient vestibular function It could be useful in the analysis of saccular and vestibulospinal tract function, detecting pathologies in inferior vestibular nerve and diagnosis of meniere's disease.saccular afferents stimulate VEMP response and this disease in early stages,affects saccular function, so this is clear that the altered saccule has different function and will cause changes in VEMP test results

ELIGIBILITY:
Inclusion Criteria:

* their age range from (25-50) years old .
* Both sexes will be included.
* Total coverage of patients attending the clinic in the fixed chosen day weekly suffering from Hypothyroidism patients with vertigo clinical diagnosis of Alzheimer's disease

Exclusion Criteria:

evidence of systemic illness except thyroid hypo function evidence of other autoimmune diseases history of head trauma neck stiffness conductive hearing loss insulin dependent diabetes

.

Ages: 25 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Study group will include 50 patients, their ages from 20 to 50 years old described with hypothyroidism.
  50 patients will be divided in to 2 groups: 1-25 patients controlled on medical treatment. 2-25 patients uncontrolled on medical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Early detection of endolymphtic hydrops in hypothyroid patients | Baseline
  Cervical vestibular evoked myogenic potential

CONTACTS AND LOCATIONS:
Overall Officials: Enas Mostafa Osman, lecturer, Study Chair — audiovestibular medicine, assiut university; mohamed salama bakr, professor, Study Director — audiovestibular medicine, assiut university

REFERENCES:
- [Background] 1. Elmoazen DM, Sobhy OA, Abd Elbaky F. Vestibular evoked myogenic potentials and video head impulse tests in different stages of Meniere's disease. Advanced Arab Academy of Audio-Vestibulogy Journal. 2015;2(2):45. 2. Baloh R, Honrubia V. Endolymphatic hydrops (Meniere's syndrome). Clinical neurophysiology of the vestibular system, 3rd ed. New York: Oxford …; 2001. 3. Friedman RA, Ryan AF. The molecular mechanism and genetics of Meniere disease. Meniere's disease: Kugler Pubblications The Hague; 1999. p. 356-69. 4. Yoo T, Ge X, Sener O, Mora M, Kwon SS, Mora F, et al. Presence of autoantibodies in the sera of Meniere's disease. Annals of Otology, Rhinology & Laryngology. 2001;110(5):425-9. 5. Fisher LM, Derebery MJ, Friedman RA. Oral steroid treatment for hearing improvement in Ménière's disease and endolymphatic hydrops. Otology & Neurotology. 2012;33(9):1685-91. 6. Hsu L, Zhu X-N, Zhao Y-S. Immunoglobulin E and circulating immune complexes in endolymphatic hydrops. Annals of Otology, Rhinology & Laryngology. 1990;99(7):535-8. 7. Garcia-Purrinos F, Ferri E, Rosell A, Calvo J. Combined intratympanic and intravenous dexomethasone to control vertigo in Meniere disease. Acta otorrinolaringologica espanola. 2005;56(2):74-7. 8. Shea JJ. Autoimmune sensorineural hearing loss as an aggravating factor in Meniere's disease. Neurophysiological and Clinical Aspects of Vestibular Disorders. 30: Karger Publishers; 1983. p. 254-7. 9. Xenellis J, Morrison A, McClowskey D, Festenstein H. HLA antigens in the pathogenesis of Meniere's disease. The Journal of Laryngology & Otology. 1986;100(1):21-4. 10. Duntas LH, Mantzou E, Koutras DA. Circulating levels of oxidized low-density lipoprotein in overt and mild hypothyroidism. Thyroid. 2002;12(11):1003-7. 11. Goebel JA. 2015 Equilibrium Committee amendment to the 1995 AAO-HNS guidelines for the definition of Meniere's disease. Otolaryngology--Head and Neck Surgery. 2016;154(3):403-4. 12. Kim C-H, Shin JE, Yoo MH, Park HJ. Direction-changing and direction-fixed positional nystagmus in patients with vestibular neuritis and meniere disease. Clinical and Experimental Otorhinolaryngology. 2019;12(3):255. 13. Alexander TH, Harris JP. Current epidemiology of Meniere's syndrome. Otolaryngologic Clinics of North America. 2010;43(5):965-70. 14. Shambaugh Jr GE. Endocrine aspects of meniere's disease. The Laryngoscope. 1959;69(8):1027-32. 15. Powers WH. Metabolic aspects of Meniere's disease. The Laryngoscope. 1978;88(1):122-9. 16. Kinney SE. The metabolic evaluation in Meniere's disease. Otolaryngology-Head and Neck Surgery. 1980;88(5):594-8. 17. Meyerhoff WL, Paparella MM, Gudbrandsson FK. Clinical evaluation of Meniere's disease. The Laryngoscope. 1981;91(10):1663-8. 18. Evans K, Baldwin D, Bainbridge D, Morrison A. Immune status in patients with Meniere's disease. Archives of oto-rhino-laryngology. 1988;245(5):287-92. 19. Seo T, Node M, Yukimasa A, Sakagami M. Furosemide loading vestibular evoked myogenic potential for unilateral Ménière's disease. Otology & neurotology. 2003;24(2):283-8. 20. Colebatch J, Halmagyi G. Vestibular evoked potentials in human neck muscles before and after unilateral vestibular deafferentation. Neurology. 1992;42(8):1635-. 21. Halmagyi G, Colebatch J, Curthoys I. New tests of vestibular function. Bailliere's clinical neurology. 1994;3(3):485-500. 22. Jacobson G. mccaslin DL. The Vestibular-Evoked Myogenic Potential and Other Sonomotor Evoked Potentials. Auditory Evoked Potentials Basic Principles and Clinical Application. USA Lippincott Williams & Wilkins. 2007;8(27):572-98. 23. Jacobson G, McCaslin D. The vestibular evoked myogenic potential and other sonomotor evoked potentials. Lippincott Williams & Wilkins Baltimore, Md, USA; 2007. p. 572-98.